CLINICAL TRIAL: NCT05592002
Title: A Multicenter Study to Assess the Safety and Effectiveness of the Genio® Dual-sided Hypoglossal Nerve Stimulation System for the Treatment of Obstructive Sleep Apnea in Subjects With Complete Concentric Collapse of the Soft Palate.
Brief Title: Safety and Effectiveness of the Genio® bilAteral Stimulation for Treatment of Complete Concentric CollapsE and OSA.
Acronym: ACCCESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nyxoah S.A. (Industry)
Collaborators: Nyxoah Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-CCC2022
Record Dates: First submitted 2022-10-13; First posted 2022-10-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Genio® 2.1 System (Experimental): System Component Genio® System 2.1 Implantable Stimulator (IS) Genio® Implantable Stimulator External Stimulator (ES) Genio® External Stimulator Disposable Patch (DP) Genio® Disposable Patch Activation Chip (AC) Genio® Activation Chip (AC) Model #2364 Charging Unit (CU) Genio® Charging Unit (CU) Model #2238 Sleep Lab Application Genio® Sleep Lab Application Smartphone Application (optional) Genio® Smartphone Application
  Interventions: Device: Genio System

INTERVENTIONS:
Device: Genio System — The Genio® IS electrode placement does not require an extensive surgical manipulation of the hypoglossal nerve, it requires only a single incision site and does not require battery replacements as those are external components. Whereas UPPP surgery and other similar upper airway enlargement surgeries are much more extensive, are irreversible and tend to have more complications and modest long-term results in reducing OSA severity and symptoms. In summary, the solution offered by the Genio System to treat OSA patients with CCC using bilateral HGNS has a favorable risk-benefit ratio, as demonstrated by evidence from 2 studies.
  Other Names: Genio System 2.0

SUMMARY:
The solution offered by the Genio System to treat OSA patients with CCC using bilateral HGNS has a favorable risk-benefit ratio, as demonstrated by evidence from 2 studies.

DETAILED DESCRIPTION:
Nyxoah has developed the Genio® 2.1 System with the intention of treating patients with moderate to severe obstructive sleep apnea.

In overview, the System includes an Implantable Stimulator (IS) designed to stimulate the hypoglossal nerve branches (i.e., both the left and the right). The IS does not include a battery but receives energy pulses transmitted by an Activation Chip (AC) which is attached to an adhesive Disposable Patch (DP) and placed on the patient's skin under the chin. Stimulation of the hypoglossal nerve causes the tongue muscles to contract with the intention to maintain an open airway.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age from 22 to 75 years (inclusive). Participant cannot be under guardianship, under curatorship or under judicial protection.

  2. Body mass index (BMI) ≤ 32 kg/m2. 3. Positive cricomental space (≥ 0 cm). The cricomental space is the distance between the neck and the bisection of a line from the chin to the cricoid membrane when the head is in a neutral position.

  4. Has either not tolerated, has failed or refused positive airway pressure (PAP) treatments.

  5. Moderate to severe OSA (15≤AHI4≤65 where combined central and mixed AHI<25% of the total AHI) based on a screening HST and confirmed in Baseline PSG.

  6. Complete concentric collapse at the level of the soft palate based on screening DISE.

  7. Willing and capable of complying with all study requirements, including specific lifestyle considerations, performing all follow-up visits and sleep studies, evaluation procedures and questionnaires for the whole duration of the trial.
* Exclusion Criteria:

  1. Inadequately treated sleep disorders other than OSA that would confound functional sleep assessment:

     1. Severe chronic insomnia,
     2. Insufficient sleep syndrome (<6 hours sleep per night),
     3. Narcolepsy,
     4. Restless legs syndrome,
     5. REM behavior disorder,
     6. Others deemed sufficient disorders that would confound functional sleep assessment in the judgment of the investigator.
  2. Taking medications that may alter consciousness, the pattern of respiration, or sleep architecture as determined by the investigator.
  3. Major anatomical or functional abnormalities that would impair the ability of the Genio® System to treat OSA:

     1. Craniofacial abnormalities narrowing the airway or the implantation site,
     2. Palatine tonsil size 3+ or 4+ by the Brodsky Classification,
     3. Fixed upper airway obstructions (tumor, polyps, nasal obstruction),
     4. Congenital malformations in the airway,
     5. Hypoglossal nerve palsy (bilateral limited tongue movement, or unilateral unintended tongue deviation during protrusion),
     6. Existing swallowing difficulty as measured by a score of ≥3 on the EAT-10 questionnaire
     7. Others deemed sufficient to impair the ability of the Genio® System to treat OSA in the judgment of the investigator.
  4. Significant comorbidities that contraindicate surgery or general anesthesia:

     1. Revised Cardiac Risk Index Class III or IV,
     2. Persistent uncontrolled diagnosed hypertension despite medications,
     3. Coagulopathy or required anticoagulant or antiplatelet medications (such as warfarin, clopidogrel (Plavix) or similar; prophylactic aspirin not exclusionary) that cannot be safely stopped in the perioperative period, Subjects meeting any of the following criteria will be excluded from participation in this study:

  <!-- -->

  1. Inadequately treated sleep disorders other than OSA that would confound functional sleep assessment:

     1. Severe chronic insomnia,
     2. Insufficient sleep syndrome (<6 hours sleep per night),
     3. Narcolepsy,
     4. Restless legs syndrome,
     5. REM behavior disorder,
     6. Others deemed sufficient disorders that would confound functional sleep assessment in the judgment of the investigator.
  2. Taking medications that may alter consciousness, the pattern of respiration, or sleep architecture as determined by the investigator.
  3. Major anatomical or functional abnormalities that would impair the ability of the Genio® System to treat OSA:

     1. Craniofacial abnormalities narrowing the airway or the implantation site,
     2. Palatine tonsil size 3+ or 4+ by the Brodsky Classification,
     3. Fixed upper airway obstructions (tumor, polyps, nasal obstruction),
     4. Congenital malformations in the airway,
     5. Hypoglossal nerve palsy (bilateral limited tongue movement, or unilateral unintended tongue deviation during protrusion),
     6. Existing swallowing difficulty as measured by a score of ≥3 on the EAT-10 questionnaire
     7. Others deemed sufficient to impair the ability of the Genio® System to treat OSA in the judgment of the investigator.
  4. Significant comorbidities that contraindicate surgery or general anesthesia:

     1. Revised Cardiac Risk Index Class III or IV,
     2. Persistent uncontrolled diagnosed hypertension despite medications,
     3. Coagulopathy or required anticoagulant medications (such as warfarin, clopidogrel (Plavix) or similar; prophylactic aspirin not exclusionary) that cannot be safely stopped in the perioperative period,
     4. Degenerative neurological disorder (i.e., Parkinson's disease, Alzheimer's disease),
     5. Acute illness or infection,
     6. Any other chronic medical illness or condition that contraindicates a surgical procedure or general anesthesia in the judgment of the investigator.
  5. Diagnosed psychiatric disease (e.g., psychotic illness, uncontrolled major depression or acute anxiety attacks) that prevents participant compliance with the requirements of the investigational study testing,
  6. Substance or alcohol abuse history within the previous 3 years. Alcohol and substance abuse are defined as follows:

     i. Alcohol: no days with less than 3 or 4 standard drinks for women and men respectively ii. Substance: the use of any substance in an amount unapproved by the investigator or considered illegal. The drugs most commonly abused include cocaine, marijuana, heroin (or substitution treatment), prescription drugs (especially painkillers), methamphetamines, and various other illegal substances.
  7. Life expectancy of less than 12 months.
  8. Prior surgery or treatments that could compromise the effectiveness of the Genio® System:

     1. Airway cancer surgery or radiation,
     2. Mandible or maxilla surgery in the previous 5 years (not counting dental treatments),
     3. Other upper airway surgery to remove obstructions related to OSA in the previous 3 months (e.g., uvulopalatopharyngoplasty (UPPP), tonsillectomy, nasal airway surgery),
     4. Prior hypoglossal nerve stimulation device implantation.
  9. Has an Active Implantable Medical Device (AIMD) even if the device can be temporarily turned off.
  10. Participation in another clinical study with an active treatment arm.
  11. Plan to become pregnant, currently pregnant, or breastfeeding during the study period.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | The duration of the study is expected to be approximately 4.5 years.
  The effectiveness endpoint of the study is assessed through the reduction in the severity of OSA over a period of 12 months post-implant. Primary effectiveness endpoint: percentage of responders based on a change in apnea-hypopnea index (AHI4) and oxygen desaturation index (ODI4) at 12 months post-activation. A responder is defined as any subject with a reduction of 50% in AHI4 from Baseline and a remaining AHI4 < 20 events/hour (aka "Sher Criteria"), AND 25% in ODI4 from Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jey Subarroyan, PhD, Study Director — Nyxoah S.A.
Locations (16):
- United States (16):
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - ENT and Allergy Associates of Florida, LLC, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - PharmaDev Clinical Research Institute,, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Center for ENT and Allergy, PC Ascension Medical Group, Carmel, Indiana
  - University of Iowa Institute for Clinical & Translational Science, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Massachusetts Eye & Ear, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - Hospital of the University Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Department of Otolaryngology, Philadelphia, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia